CLINICAL TRIAL: NCT00224237
Title: Exploring Folk Health Practices in Latinos With Chronic Medical Conditions
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Mary E. Charlson, MD, Principal Investigator, Weill Medical College of Cornell University
Other Study IDs: 0505007876
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Hypertension; Asthma; Heart Disease; Stroke; Arthritis
Keywords: Latino patients; Health practices; Culture influences
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Asthma; Heart Diseases; Stroke; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Participants will be self-identified, adult Latino men and women from the community setting. The sample will comprise of a convenience sample from community-based organizations, including persons of Mexican, Puerto Rican, Cuban, Dominican, Central American, South American, or other Spanish-speaking culture.

SUMMARY:
This study will explore how culture influences the use of folk healing practices and medical services in Latinos with chronic medical conditions.

DETAILED DESCRIPTION:
Sociocultural aspects of using ethnomedical health practices in a community-based Latino population will be described using both qualitative and quantitative survey methods. This study will rely heavily on its descriptive section, which will use in-depth, open-ended questions in a semi-structured personal interview format following qualitative research principles. It will also use closed-ended questions in a short survey format to begin to explore some variables that may be associated with using traditional healing practices. These variables include level of acculturation, degree of family social support, degree of adherence to standard medical regimens, perceived health status, presence of depressive symptoms, and severity of co-illnesses. These variables will be examined using common, validated scales.

ELIGIBILITY:
Inclusion Criteria:

Participants will be self-identified, adult men and women from the community setting. The sample comprise a convenience sample, including persons of Mexican, Puerto Rican, Cuban, Dominican, Central American, South American, or other Spanish speaking culture.

1. Latino men and women over the age of 18
2. Those self-identifying as having at least one chronic medical condition including:diabetes, hypertension, asthma, history of heart disease or stroke or musculoskeletal disease (arthritis).
3. Those reporting use of complementary or alternative therapies, including ethnomedical healing practices or practitioners.
4. Those who speak English or Spanish.

Exclusion Criteria:

Individuals who refuse to participate.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be self-identified, adult Latino men and women from the community setting. The sample will comprise of a convenience sample from community-based organizations, including persons of Mexican, Puerto Rican, Cuban, Dominican, Central American, South American, or other Spanish-speaking culture.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2005-12 (Actual); Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Duarte, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- The New York Presbyterian Hospital-Weill Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No Plan to Share IPD